CLINICAL TRIAL: NCT00237094
Title: Use of Midlevel Providers in Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65787 (completed); 1R18DK065787-01A1 (NIH)
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Self Management; Interdisciplinary team
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Behavioral: Nurse Practitioner led multidisciplinary team approach

SUMMARY:
Studies have demonstrated that intensive disease management of diabetes and its associated risk factors, hypertension and dyslipidemia, can prevent the progression of vascular complications. However, implementation of well defined guidelines for intensive disease management has been suboptimal. Barriers to success occur at multiple levels, including health care systems, health care providers and patients.

In rural regions of the U.S., reduced availability of primary care providers and specialty services, including diabetes education, present additional barriers to effective diabetes care. Use of a nurse practitioner led interdisciplinary team to intensively manage urban and rural diabetic patients, utilizing telehealth technology to provide care to rural areas, will help begin to address these barriers

The long term goal of the project is to develop a practical and sustainable system of intensive diabetes management that will be effective in helping diabetic patients achieve and maintain goals within established treatment guidelines regardless of geographic location.

Specific aims are:

1. To determine in both urban and rural areas if a nurse practitioner led team approach to intensive diabetes management and education improves disease-specific outcomes and patient education compared to traditional care (current diabetes management of urban patients).
2. To determine if telehealth is an effective and accepted mechanism for delivery of a nurse practitioner led team approach to intensive diabetes management and education in rural areas.
3. To determine if a nurse practitioner led intensive disease management team can identify patient risk factors (psychological, financial, and work-related factors) that may be barriers to patient adherence, earlier in the management of urban diabetic patients compared to traditional care.
4. To compare volume and type of service utilization of a nurse practitioner led team approach to diabetes management and education to that of traditional care in both urban and rural areas. Disease-specific outcomes will include physiologic variables (HbA1c, blood pressure, lipid levels), measurement and documentation of preventive services (dilated eye exam, monofilament exam, microabumin testing) and patient's knowledge of disease tested by questionnaire.

Results should show improved outcomes and patient knowledge in urban and rural patients receiving intensive disease management compared to traditional care.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of Type II diabetes based on ADA diagnostic criteria.
* All persons with diabetes who do not meet ADA goals for glycemic, blood pressure or lipid control.This includes new or previously diagnosed patients.
* Men and women 21 years of age or older.
* Speaks and reads English
* Willing to participate (informed consent)

Exclusion Criteria:

* Type I diabetes
* Diagnosis of dementia or mental retardation.
* Resident of personal care home, assisted living, or long term care facility.
* Significant drug/alcohol abuse in the past 18 months.
* Active malignant process including patients on chemotherapy.
* Steroid induced diabetes or patient on chronic or intermittent steroid therapy (use for more than 2 months out of a year)
* Acute or chronic inflammatory or infectious disease process (chronic osteomyelitis, HIV, tuberculosis, bacterial endocarditis)
* End stage renal or liver disease.
* Pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Coon, MD, Principal Investigator — Deaconess Billings Clinic
Locations (1):
- Deaconess Billings Clinic Center on Aging, Billings, Montana, United States